CLINICAL TRIAL: NCT03512938
Title: Effects of Smoking on Non-surgical Periodontal Therapy in Generalized Aggressive Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Principal Investigator, Nurcan Buduneli, Clinical Professor, Ege University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-DIS-013
Record Dates: First submitted 2018-03-24; First posted 2018-05-01 (Actual); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Generalized Aggressive Periodontitis; Smoking
Keywords: Generalized aggressive periodontitis; Non-surgical periodontal therapy; Periodontopathogens; Smoking; Gingival crevicular fluid
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-smoker Group (Active Comparator): This group included non-smoker generalized aggressive periodontitis patients.
  Interventions: Procedure: Non-surgical periodontal therapy
- Smoker Group (Experimental): This group included smoker generalized aggressive periodontitis patients.
  Interventions: Procedure: Non-surgical periodontal therapy

INTERVENTIONS:
Procedure: Non-surgical periodontal therapy — Patients were motivated and instructed to brush with modified Bass technique and use interdental toothbrushes, dental floss. Each patient underwent quadrant scaling and root planning (SRP) under local anaesthesia over a 4-week period. Root planing (RP) was performed under local anaesthesia (2% lidocaine, epinephrine 1:100.000) and a standard curette set newly sharpened with Arkansas stone was used for each patient.

SUMMARY:
Smoking is the major preventable risk factor in the initiation and progression of periodontal diseases. Periodontitis risk was found to be 3.9 times higher among smokers aged between 19-30 years and 2.8 times higher among smokers aged 31-40 years compared to non-smokers. Aggressive periodontitis (AgP), is characterized by a rapid attachment loss usually incompatible with the amount of plaque and dental calculus. It is often not possible to predict the prognosis of treatment with various treatment options in cases of aggressive periodontitis. It was hypothesized that non-smoker patients with generalized aggressive periodontitis (GAgP) will respond better to conventional mechanical non-surgical periodontal therapy compared to the smokers. Therefore, the aim of this study was to evaluate the effects of smoking on the outcomes of non-surgical periodontal treatment in terms of the clinical, biochemical and microbiological parameters.

ELIGIBILITY:
Inclusion Criteria:

* Having at least six permanent teeth, including incisors and/or first molars with severe periodontal disease
* Having at least one site with probing depth (PD) and clinical attachment level (CAL) ≥5 mm and six teeth other than first molars and incisors with similar PD and CAL measurements
* Familial aggregation

Exclusion Criteria:

* Medical disorders such as diabetes mellitus, immunological disorders
* Having an antibiotic or periodontal treatment in the last 6 months
* Having <15 teeth

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2014-06-23 (Actual); Primary Completion 2016-02-08 (Actual); Study Completion 2017-09-28 (Actual)

PRIMARY OUTCOMES:
Change in Clinical Attachment Level (CAL) | Baseline and 1 month, 3 month, 6 month after non-surgical periodontal therapy

SECONDARY OUTCOMES:
Change in Probing Depth (PD) | Baseline and 1 month, 3 month, 6 month after non-surgical periodontal therapy
Change in Bleeding on Probing (BoP) | Baseline and 1 month, 3 month, 6 month after non-surgical periodontal therapy
Change in Plaque Index (PI) | Baseline and 1 month, 3 month, 6 month after non-surgical periodontal therapy
Changing of the salivary biomarkers | Baseline and 1 month, 3 month, 6 month after non-surgical periodontal therapy
  In the morning following an overnight fast, during which subjects were requested not to drink (except water) or to chew gum, whole saliva samples were obtained by expectorating into polypropylene tubes; clinical periodontal measurements and any necessary periodontal interventions were then carried out. Cytokine levels were assessed by Enzyme-linked immunosorbent assay (ELISA).
Changing of the serum biomarkers | Baseline and 1 month, 3 month, 6 month after non-surgical periodontal therapy
  Nine milliliters of venous blood were taken from the antecubital vein by a standard venipuncture method and centrifuged for 10 minutes at 3,000 rpm, separating serum from the cells. Cytokine levels were assessed by Enzyme-linked immunosorbent assay (ELISA).
Changing of the gingival crevicular fluid (GCF) biomarkers | Baseline and 1 month, 3 month, 6 month after non-surgical periodontal therapy
  GCF samples were obtained from buccal aspects of one interproximal site in each quadrant. Supragingival plaque was removed carefully by sterile curettes; the surfaces were dried and isolated by cotton rolls. Filter paper strips were placed in the orifices of the gingival sulcus/pocket for 30 seconds. Care was used to avoid mechanical trauma, and strips contaminated with blood were discarded. The absorbed GCF volume was estimated by a calibrated instrument. The readings of GCF sample volumes were converted to an actual volume (μL) by reference to the standard curve. Cytokine levels were assessed by Enzyme-linked immunosorbent assay (ELISA).
Changing of the amount of pathogen microorganisms | Baseline and 1 month, 3 month, 6 month after non-surgical periodontal therapy
  Plaque samples were collected from the same sites by sterile paper points from the base of the pockets. Paper points were inserted into the deepest part of the pocket and kept for 5 seconds. Paper points were then placed into propylene tubes. Real-time polymerase chain reaction was used for detection and quantification of bacterial cell copy numbers in 1 mg plaque.